CLINICAL TRIAL: NCT01920581
Title: Assessment of Problematic Use of Benzodiazepines and Z Drugs in the Elderly in France: a Public Health Issue
Brief Title: Use of Benzodiazepines and Z Drugs in the Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/10/06-W
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Benzodiazepines and Related Drugs Users
Keywords: CEIP; pharmacodependance; addictovigilance; benzodiazepines and benzodiazepines related drugs; elderly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- volunteers

SUMMARY:
The aim of this study is to evaluate benzodiazepines and related drugs (zolpidem and zopiclone) usage in an outpatient population of chronic users over 65 years in France using a questionnaire assessing substance dependence according to DSM-IV (Diagnostic and Statistical Manual of mental disorders) international standards.

DETAILED DESCRIPTION:
1100 patients will be recruited by pharmacists. They will answer to a standardized questionnaire assessing their benzodiazepines or related drugs usage (phone contact).

Pharmacists are recruited by all French Centers For Evaluation and Information on Pharmacodependence (CEIP).

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or more,
* benzodiazepines or benzodiazepines related drugs treatment for at least three months,
* written consent and without exclusion criteria.

Exclusion Criteria:

* no written consent form
* difficulties to understand or speak french

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 65 years old or more volunteers,with benzodiazepines or benzodiazepines related drugs treatment for at least three months, written consent and without exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Dependence according to DSM IV criteria | 2 years

SECONDARY OUTCOMES:
withdrawal syndrome | 2 years
psychiatric comorbidities | 2 years
Dependence scores | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Jolliet, PUPH, Study Director — Nantes University Hospital
Locations (11):
- France (11):
  - CEIP Bordeaux, Bordeaux
  - CEIP Caen, Caen
  - CEIP Grenoble, Grenoble
  - CEIP Lille, Lille
  - CEIP Lyon, Lyon
  - CEIP Marseille, Marseille
  - CEIP Montpellier, Montpellier
  - CEIP Nancy, Nancy
  - CEIP Nantes, Nantes
  - CEIP Paris, Paris
  - CEIP Toulouse, Toulouse

REFERENCES:
- [Derived] Victorri-Vigneau C, Laforgue EJ, Grall-Bronnec M, Guillou-Landreat M, Rousselet M, Guerlais M; FAN-Network; Feuillet F, Jolliet P. Are Seniors Dependent on Benzodiazepines? A National Clinical Survey of Substance Use Disorder. Clin Pharmacol Ther. 2021 Feb;109(2):528-535. doi: 10.1002/cpt.2025. Epub 2020 Sep 23. PMID 32860424